CLINICAL TRIAL: NCT00017498
Title: Phase II Study On Gemcitabine In Recurrent Or Metastatic Adenoid Cystic Carcinoma Of The Head And Neck
Brief Title: Gemcitabine in Treating Patients With Recurrent or Metastatic Adenoid Cystic Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-24982; EORTC-24982
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: stage IV salivary gland cancer; recurrent salivary gland cancer; salivary gland adenoid cystic carcinoma; stage IV adenoid cystic carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating patients who have recurrent or metastatic adenoid cystic cancer of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the therapeutic activity of gemcitabine, in terms of objective response and duration of response, in patients with recurrent or metastatic adenoid cystic carcinoma of the head and neck.
* Determine the acute toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30-60 minutes on days 1 and 8. Treatment repeats every 21 days for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 12 weeks until disease progression and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 16-29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or recurrent adenoid cystic carcinoma of the head and neck for which no curative options exist

  * Symptomatic and/or progressive disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * No bone metastases as only lesion
  * Prior radiotherapy to only target lesion allowed if it has progressed or reappeared after radiotherapy
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN) (2.5 times ULN if liver metastases present)
* AST or ALT less than 3 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.7 mg/dL

Other:

* No uncontrolled infection
* No concurrent serious systemic disorders that would preclude study
* No other prior or concurrent malignancy except:

  * Adequately treated carcinoma in situ of the cervix
  * Basal cell or squamous cell skin cancer
  * Any malignancy that occurred more than 5 years ago with no symptoms or signs of recurrence (except malignant melanoma, hypernephroma, or breast carcinoma)
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent anti-estrogen therapy
* Concurrent steroid replacement or steroids as an antiemetic allowed

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy except for palliative radiotherapy to bone lesions
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 1 month since prior investigational agents
* No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-02; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter H. M. de Mulder, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (7):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Italy (2):
  - Ospedale Santa Croce, Cuneo
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - University Medical Center Nijmegen, Nijmegen

REFERENCES:
- [Result] van Herpen CM, Locati LD, Buter J, Thomas J, Bogaerts J, Lacombe D, de Mulder P, Awada A, Licitra L, Bernier J, Vermorken JB. Phase II study on gemcitabine in recurrent and/or metastatic adenoid cystic carcinoma of the head and neck (EORTC 24982). Eur J Cancer. 2008 Nov;44(17):2542-5. doi: 10.1016/j.ejca.2008.08.014. Epub 2008 Sep 24. PMID 18819792